CLINICAL TRIAL: NCT01366508
Title: An Experimental Medicine Study to Characterize Event Related Potential Markers of Attentional Bias Towards Words and Images of Food in Healthy Volunteers
Brief Title: A Study to Characterize Event Related Potential Markers of Attentional Bias Towards Words and Images of Food
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Results of the study would unfortunately no longer be of any scientific interest to the sponsor and would not be used to inform future studies.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 112336
Record Dates: First submitted 2011-04-14; First posted 2011-06-06 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Breakfast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visit B (Other): At approximately 09:00 the subject will be given breakfast. After this, no food will be served until study procedures for the day are over. However, a 330 ml bottle of still water at room temperature will be given at ~11:00 and at ~13:00. During this period the subject will be required to remain in the unit.
  Interventions: Other: High calorie lunch; Other: Breakfast
- Visit A (Other): At approximately 13:00 the subject will be given a standard high calorie lunch that the subject is required to finish
  Interventions: Other: High calorie lunch; Other: Breakfast

INTERVENTIONS:
Other: High calorie lunch — Subject fed a standard high calorie lunch at 1pm
Other: Breakfast — At approximately 09:00 the subject will be given breakfast. After this, no food will be served until study procedures for the day are over. However, a 330 ml bottle of still water at room temperature will be given at ~11:00 and at ~13:00. During this period the subject will be required to remain in the unit.

SUMMARY:
GSK is planning to undertake two anti-obesity drug studies in the area of obesity. In addition to assessment by questionnaires, it would be of significant value to incorporate an objective non-interventional measure of cognitive or motivational processing associated with evaluating and responding to food stimuli. Obesity is associated with increased attentional bias to palatable foods. The aims of this protocol are two-fold, first to characterize Event Related Potentials (ERPs) of two common aspects of food stimuli relevant to eating disorders -presence of food and its palatability, and secondly, to assess the modulation of these ERPs by appetite. Following a successful completion of this study, it is the intention to use the paradigm developed in future studies in the area of obesity.

DETAILED DESCRIPTION:
GlaxoSmithKline is currently developing a number of drugs for the treatment of overheating including 'binge eating' in obesity. Historically, the behavioural effectiveness of anti-obesity drugs in clinical drug trials have utilised subjective rating scales to assess a person's drive or motivation to eat. Findings from these studies have good construct validity, but suffer from the shortcomings of self-reporting, e.g. the subject bias, dishonesty, misinterpretation. It follows that in addition to self-reporting, it would strengthen the interpretation of any future studies on anti-obesity drugs, if there were to be an objective measure of brain activity in relation to cognitive/motivational processes associated with evaluation and responding to food related cues.

Measuring event related potentials (ERPs) during cognitive processes of food related cues, using the electroencephalography technique (EEG) offers a an alternative objective approach to examining the effectives of anti-obesity drugs.

This protocol proposes to develop and use two cognitive tasks examining response to food related cues (pictorial and words) with concurrent recording of ERPs, in order to characterize neurophysiological events associated with attentional bias towards food related stimuli.

The first task is an image processing task. This task uses food images similar to those in the International Affective Picture System (IAPS) used in ERP studies of perceptual processing of emotional stimuli [Olofsson, 2008; Schupp, 2006]. In this task a subject views different categories of images; palatable high-calorie food images, non-palatable low-calorie food images and non-edible plant images. The latter is the neutral category against which the ERPs of the two food categories will be compared. Affective pictures have been used to assess emotional valence by measuring differences in anterior ERP measurements between images from differing groups.

The protocol also proposes to measure late positive potential in order to assess higher level cognitive processing possibly with early memory formation. Again, the proposal is to assess AUCs, in this case in the 400-600 ms region and then look at difference curves between the late potential potentials to different valency stimuli. For the late positive potentials, anterior laterality will also be assessed. The second task is a cued-target task of visuospatial attention to motivationally salient words. The task is a version of the Posner paradigm. The appearance of a food or nonfood word inside a top or bottom frame (the cue) distracts the attention of the subject towards that spatial location. Following the word either one of the two frames changes appearance (the target).

In addition to these emotion and attention measures, the protocol proposes to assess the more standard N1, P1 and P3 [Luck, 2005]. After completing the ERP recordings the subject will be asked to rate each picture for salience and valence in order to provide a comparison between objective neurophysiological and subjective attention and emotional ratings.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as judged by the responsible physician or designee based on a medical evaluation including medical history.

  1. Right handed male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
  2. BMI within the range 27 - 35 kg/m2 (inclusive).
  3. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

  1. The subject has either a previous disease or current medical condition, which as judged by the Investigator, may affect the interpretation of efficacy data. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematological disease, neurological disease, psychiatric diseases or endocrine disease.
  2. The subject has a positive urine drug screen. A minimum list of drugs that will be screened for include Amphetamines, Barbiturates, Cocaine, Opiates, Cannabinoids, Methadone and Benzodiazepines.
  3. The subject has a history of alcohol or substance abuse or dependence in the 6 months prior to screening as determined by the investigator. Abuse of alcohol, defined for males, as an average weekly intake of greater than 28 units (or an average daily intake of greater than 4 units). One unit is equivalent to a half-pint (220mL) of beer or 1 (25mL) measure of spirits or 1 glass (125mL) of wine.
  4. A positive alcohol breath test.
  5. The subject has a history of stroke, seizures, epilepsy or abnormal EEG.
  6. The subject is a smoker.
  7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
  8. Subjects who are currently taking any regular medication.
  9. Subject has a history of clinically significant eating disorders.
  10. Subject is a vegetarian.
  11. Subject is a member of GlaxoSmithKline Clinical Unit staff.
  12. Subject is female.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Event Related Potential Amplitude, Latency and Area Under the Curve, Reaction | 1 hour

SECONDARY OUTCOMES:
Hip-to-waist ratio and BMI | 6 hours

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, United Kingdom